CLINICAL TRIAL: NCT06317701
Title: Hgns: Metabolic Endpoints For Obstructive Sleep Apnea Following Twelfth Cranial Nerve Stimulation
Brief Title: Metabolic Endpoints for Obstructive Sleep Apnea Following Twelfth Cranial Nerve Stimulation
Status: Recruiting | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: IRB23-1801
Record Dates: First submitted 2024-02-28; First posted 2024-03-19 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- HGNS Therapy Participants: Individuals with sleep apnea treated by HGNS therapy.
  Interventions: Device: Hypoglossal Nerve Stimulation (HGNS)
- patients with OSA and complete concentric airway collapse on DISE: By standard of care, patients undergoing evaluation for HGNS as an alternative therapy for OSA must undergo drug-induced sleep endoscopy (DISE) to confirm anterior-posterior airway collapse (APC) and rule out complete concentric airway collapse (CCC). Currently, no studies have described the cardiometabolic profiles of patients with OSA and CCC - a population that is both intolerant to PAP and ineligible for HGNS.
  participants with CCC on DISE will complete an identical set of measures as the APC group. Due to the presence of CCC, these participants will not undergo surgery and will only receive testing once. Data from these subjects will be compared against the baseline (pre-operative) data of the APC group.

INTERVENTIONS:
Device: Hypoglossal Nerve Stimulation (HGNS) — Alternative therapy for Obstructive Sleep Apnea
  Groups: HGNS Therapy Participants

SUMMARY:
The purpose of this study is to determine if the treatment of Obstructive sleep apnea (OSA) by hypoglossal nerve stimulation (HGNS) will alter glucose metabolism. The study team will also determine if the treatment of Obstructive sleep apnea (OSA) by (hypoglossal nerve stimulation) HGNS will alter predictors of cardiovascular outcomes.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a highly prevalent sleep disorder in the general population. It is estimated that 80 percent of those who have OSA remain undiagnosed, and thus do not receive therapy. Strong evidence from epidemiologic and clinical studies suggests that untreated OSA is an independent risk factor for cardiometabolic disease, particularly among those with moderate-to-severe OSA. Animal and human models have revealed that intermittent hypoxia and sleep fragmentation (i.e., main features of OSA) result in insulin resistance, glucose intolerance and pancreatic beta-cell dysfunction, hypertension and dyslipidemia. Continuous positive airway pressure (CPAP) is the established first-line treatment for OSA. However, only 50% of patients with OSA are adherent to CPAP therapy. Notably, a key limitation of prior CPAP trials on cardiometabolic outcomes is low treatment adherence.

A randomized controlled trial conducted at the University of Chicago demonstrated that 8 hours of nightly CPAP reduces glucose response during oral glucose tolerance testing and improves insulin sensitivity in individuals with OSA and prediabetes. In 2014, following the pivotal Safe and Timely Antithrombotic Removal - Ticagrelor trial (STAR), the Food and Drug Administration (FDA) approved hypoglossal nerve stimulation (HNS) as an alternative therapy for OSA. Five-year outcomes from STAR have confirmed durable efficacy, tolerance, and safety for HNS. From improved tolerance and adherence, it is theorized that HNS may be more effective than CPAP at ameliorating cardiovascular and diabetes risk. Yet, there is no literature on the cardiometabolic outcomes of treating OSA with HNS.

The study team's long-term goal is to understand the metabolic and cardiovascular effects of OSA and how current therapies can mitigate risk and improve outcomes. The overall objective of this study is to determine the cardiometabolic impact of HNS therapy in patients with moderate-to-severe OSA who are intolerant to CPAP. It is hypothesized by the investigator that effective HNS treatment will improve glucose metabolism and markers of cardiovascular disease.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese males and females BMI 25 kg/m2 to 40 kg/m2
* Age 18 years and older
* Diagnosed with obstructive sleep apnea by Apnea-Hypopnea Index >15 events/hr using 4% oxygen desaturation criteria and < 25% central events/hr on prior sleep testing Data can be derived from home sleep testing or in-lab polysomnogram
* Not able to use positive airway pressure >4 hours for 5 nights/week or unwilling to use positive airway pressure

Exclusion Criteria:

* Insulin-dependent Diabetes
* Inability to undergo in-lab polysomnography or home sleep testing
* Central Nervous System (CNS) disease with impairment of cognitive function (dementia) and/or muscle paresis, such as stroke
* Currently pregnant, trying to get pregnant or nursing
* age < 18 years
* Regular and adherent CPAP use per clinical guidelines
* Current night shift or rotating shift work
* Diagnosis of another sleep disorder (e.g. periodic limb movement disorder)
* Current systemic steroid use
* Predominantly central sleep apnea or requiring oxygen or bi-level positive airway pressure or advanced positive airway pressure modalities
* Protected patient: under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision, including hospitalized without consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects will be recruited from the Sleep Surgery Clinic of the Duchossois Center for Advanced Medicine (DCAM) in Hyde Park and Sleep Surgery Clinic of UChicago Medicine - Orland Park and Hinsdale.. We will take advantage of the electronic medical records (EMR) to identify potential candidates using databases (EPIC-based) from the University of Chicago and Ingalls. Participants will be identified by an initial screening of patients scheduled in EPIC for drug induced sleep endoscopy (DISE).
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Glycemic variability | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-op
  measured by standard deviation (SD) of average blood glucose or % coefficient of variation (SD / mean glucose) on two-week continuous glucose monitor
Mean systolic BP (daytime and nocturnal) | 24 hrs at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-op
  important mediators of cardiovascular outcomes
Glycemic variability | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-op
  measured by standard deviation (SD) of % coefficient of variation (SD / mean glucose) on two-week continuous glucose monitor

SECONDARY OUTCOMES:
mean blood glucose levels | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
  other glycemic metrics for the clinical care of diabetes to be followed.
mean ambulatory glucose excursions | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
  glycemic metrics for the clinical care of diabetes will be followed
time blocks | 24-h, day, night at baseline and after HGNS implant, acclimation, and tuning
  glycemic metrics for the clinical care of diabetes will be followed
Morning fasting insulin, including calculated insulin resistance (HOMA-IR) | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
Mean norepinephrine levels | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
Morning fasting blood glucose | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
  markers of glucose metabolism
Hemoglobin A1c | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
  markers of glucose metabolism
Insulin levels | at baseline and after HGNS implant, acclimation, and tuning
  markers of glucose metabolism
c-peptide levels | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
  markers of glucose metabolism
fasting lipid profile (triglycerides) | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
  testing for signs of cardiovascular disease
heart rate indices by activity monitor | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
  testing for signs of cardiovascular disease
sympathetic activity by plasma norepinephrine | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
  to investigate its role as a mediator in cardiometabolic response to treatment
Morning fasting insulin of c-peptide level | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
fasting lipid profile (HDL- cholesterol) | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
  testing for signs of cardiovascular disease
fasting lipid profile ( LDL-cholesterol) | at baseline and after HGNS implant, acclimation, and tuning at 3 month Post-Op
  testing for signs of cardiovascular disease

CONTACTS AND LOCATIONS:
Overall Officials: Phillip LoSavio, MD, MS, Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No